CLINICAL TRIAL: NCT06344013
Title: The ABCDEF Bundle in Critical Care: a French National Survey Still a Long Way to go!
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0034 - BUNDLE ABCDEF
Record Dates: First submitted 2024-03-26; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Delirium
Keywords: ABCDEF bundle, ICU delirium, sedation, exercise, family
MeSH Terms: conditions — Delirium; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the knowledge and compliance of French intensive care units with the ABCDEF (A: Assessment, Prevention, Management of Pain, B: Both Spontaneous Awakening Trials and Spontaneous Breathing Trials, C: Choice of Sedation and Analgesia, D: Delirium Assessment, Prevention, and Management, E: Early Mobility and Exercise, F: Family Engagement and Empowerment) bundle. French ICU doctors will be asked to answer a questionnaire available online.

ELIGIBILITY:
Inclusion Criteria:

French ICU doctors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: French ICU doctors
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
knowledge and compliance of French intensive care units with the ABCDEF | one-time evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement